CLINICAL TRIAL: NCT01080066
Title: A Post Marketing Surveillance Study of Cetuximab in Patients With Squamous Cell Carcinoma of Head and Neck (SCCHN)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Choice Pharma Taiwan (Unknown)
Responsible Party: Sponsor
Other Study IDs: EMR62202-512
Record Dates: First submitted 2010-02-18; First posted 2010-03-03 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Carcinoma; Squamous cell; Erbitux; cetuximab; Head; Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Interventional Study
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Subjects administered with Cetuximab, once weekly by intravenous infusion at a first dose of 400 milligram per square meter (mg/m^2) body surface area for 120 minutes infusion period and subsequently at a dose of 250 mg/m^2 for 60 minutes infusion period, will be observed. The maximum infusion rate must not exceed 10 milligram per minute (mg/min).
  Other Names: Erbitux®

SUMMARY:
This is a prospective, observational, non-interventional, multicenter, post-marketing surveillance study to mainly collect safety information from subjects with locally advanced and recurrent/metastatic Squamous Cell Carcinoma of Head and Neck (SCCHN) treated with cetuximab based on the locally approved label.

DETAILED DESCRIPTION:
Cetuximab is an immunoglobulin G1 (IgG1) monoclonal antibody that enhances the effects of some common chemotherapy agents and radiotherapy and demonstrates minimal overlapping toxicities with these approaches. This prospective, observational, non-interventional and multi-centric post marketing surveillance study is being conducted to collect safety information from subjects with locally advanced or recurrent/metastatic SCCHN treated with cetuximab based on the locally approved label. Study plans to enroll 200 to 300 subjects, who are eligible for cetuximab treatment according to the indication in the approved label of cetuximab by Taiwan Health Authority. Data related to subjects' demographics, relevant tumor history, and laboratory information (hematology, biochemistry) will be captured and analyzed descriptively.

OBJECTIVES

Primary objective:

• To obtain safety information on the use of cetuximab in subjects with SCCHN according to the regulatory approved label and in a regular clinical setting

Secondary objectives:

• To gather clinical efficacy information of the treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Stage 3-4 locally advanced SCCHN (oropharynx, hypopharynx, larynx) or recurrent and/or metastatic SCCHN
* Age greater than or equal to 18 years
* Signed informed consent

Exclusion Criteria:

* Subjects with known severe (Grade 3 or 4; National Cancer Institute Common Toxicity Criteria Version 4.03) hypersensitivity reactions to Cetuximab
* Subjects with contraindications for concomitantly used chemotherapeutic agents or radiation therapy, identified before initiation of cetuximab combination treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with SCCHN and are eligible to receive cetuximab and radiotherapy according to the local label
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reactions and serious adverse drug reactions | From the first infusion of cetuximab until three months after the last infusion of Cetuximab
Number of subjects discontinuing the study due to intolerability of cetuximab | From the first infusion of cetuximab until three months after the last infusion of Cetuximab

SECONDARY OUTCOMES:
Number of subjects with best tumor response categories that are, complete response, partial response, stable disease, progressive disease and not evaluable | From the first infusion of cetuximab until three months after the last infusion of cetuximab
Time to progression | From the first infusion of cetuximab until three months after the last infusion of cetuximab
Duration of response | From the first infusion of cetuximab until three months after the last infusion of cetuximab
Overall Survival | From the first infusion of cetuximab to death until three months after the last infusion of cetuximab

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Jung Tsao, Dr., Principal Investigator — Liouying Chi-Mei Hospital
Locations (1):
- Liouying Chi-Mei Hospital, Liuying, Tainan County, Taiwan